CLINICAL TRIAL: NCT01383876
Title: Collar Immobilization Following a Posterior Cervical Laminectomy and Fusion: A Randomized Controlled Trial
Brief Title: Collar Immobilization Following a Posterior Cervical Laminectomy and Fusion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment too slow
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Christopher Bono, Christopher M. Bono, MD, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010P002931
Record Dates: First submitted 2011-06-27; First posted 2011-06-28 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Cervical Spondylosis Symptomatic Neurological Compression
Keywords: cervical; laminectomy; fusion; neurological compression; spondylosis
MeSH Terms: conditions — Spondylosis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Collar (Active Comparator): Hard cervical collar placed in the operating room after surgery. The collar will be removed/exchanged for bathing, grooming, and dressing changes only. It will remain in place for 12 weeks.
  Interventions: Behavioral: Collar
- No Collar (Experimental): Have a hard cervical collar placed in the operating room after surgery. This will remain in place for 1 to 2 days and be discontinued prior to discharge.
  Interventions: Behavioral: No Collar

INTERVENTIONS:
Behavioral: Collar — Have a hard cervical collar placed in the operating room after surgery. The collar will be removed/exchanged for bathing, grooming, and dressing changes only. It will remain in place for 12 weeks.
  Arms: Collar
Behavioral: No Collar — Have a hard cervical collar placed in the operating room after surgery. This will remain in place for 1 to 2 days and be discontinued prior to discharge.
  Arms: No Collar

SUMMARY:
Cervical collars are commonly used to provide external immobilization after elective Posterior Cervical Laminectomy and Interbody Fusion (PCLIF). The rationale for collar use is the perception and assumption that it can prevent early instrumentation failure and promote successful spinal fusion. However, there are a number of potential complications associated with cervical collars such as skin breakdown, ulceration, neck pain, impedance upon activities of daily living, and impaired swallowing. Considering these conflicting factors, there is wide disagreement among spinal surgeons about the utility, benefits, and necessity of collar use following elective PCLIF.

Hypothesis: Wearing a cervical collar for 12 weeks after posterior cervical laminectomy and instrumented fusion will not demonstrate substantial benefits as measured by the incidence of instrumentation failure, rate of nonunion, or clinical outcome measures.

Specific Aim I: To compare the outcomes of surgery in patients who will wear a cervical collar for 12 weeks following surgery versus those who will have the collar removed prior to discharge after surgery.

DETAILED DESCRIPTION:
Following the informed consent process, subjects will fill out a baseline questionnaire consisting of demographic information, visual analog scale (VAS) pain scores for neck and arm pain, and the Neck Disability Index Questionnaire (NDI).

Following surgery, the surgeon will fill out an operative data collection sheet to record information such as: levels fused, type of instrumentation, pre- and post-operative sagittal alignment, and intra-operative complications (if applicable). Subjects will be randomized into the "collar" or "no collar" group immediately following surgery, using a computer generated randomization scheme, so as not to influence the surgeon's operative technique. If the patient is randomized to the "no collar" group, he or she will actually have a hard cervical collar placed in the operating room after surgery. This will remain in place for 1 to 2 days and be discontinued prior to discharge. If the patient is randomized to the "collar" group, he or she will have the hard cervical collar placed after surgery. The collar will be removed/exchanged for bathing, grooming, and dressing changes only. It will remain in place for 12 weeks.

The patient will undergo usual and customary clinical and radiographic follow-up. This includes physical examination and cervical radiographs taken at 2 weeks, 12 weeks, 6 month, and 1 year. VAS and Neck Disability Index scores will be obtained at the 2 week, 12 week, 6 month, and 1 year follow-up visits. Radiographs will be assessed by a two independent radiologists for instrumentation failure (defined as any of the following: screw loosening, screw breakage, rod breakage, screw dislodgement) and fusion status. Solid fusion will be defined as bridging trabecular bone between or along the lateral masses/facet joints of the operated segments as assessed on a lateral cervical radiograph. In addition, the overall sagittal alignment of the spine will be measured. For the primary outcome of the study, final follow-up at 1 year would be considered satisfactory to determine differences in pseudarthrosis and instrumentation failure.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* English Speaking
* Diagnosis of degenerative cervical spondylosis with symptomatic neurological compression (spinal cord and/or nerve root) requiring posterior decompression and instrumentation fusion
* Surgical construct to include instrumentation and fusion as proximal as C2 and as distal as T2
* Ability to provide written consent
* Ability to complete pre- and postoperative questionnaires

Exclusion Criteria:

* Diagnosis of malignancy, infection, fracture/dislocation of the cervical spine
* Posterior cervical constructs including the occiput or C1
* Previous cervical fusion to the occiput or C1
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2011-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Fusion Rates | 1 year
  To compare the solid fusion rates between collar and no collar groups.

SECONDARY OUTCOMES:
Clinical Outcomes | 1 year
  VAS and Neck Disability Index scores will be used to assess the clinical outcomes of both the collar and no collar groups.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Bono, M.D., Principal Investigator — Brigham & Women's Hospital, Harvard Medical School; Dana A Leonard, B.A., Study Director — Brigham and Women's Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts